CLINICAL TRIAL: NCT06708234
Title: Frequency of Isthmocele Following Single- Vs Double-layer Uterine Closure. a Prospective and Retrospective Multicenter Observational Study
Brief Title: Frequency of Isthmocele Following Single- Vs Double-layer Uterine Closure.
Status: Recruiting | Type: Observational
Sponsor: Lorenza Driul (Other)
Responsible Party: Sponsor-Investigator, Lorenza Driul, Principal investigator, Head of the Clinic Gynecology and Obstetrics Clinic, University of Udine
Organization: University of Udine (Other)
Other Study IDs: 154230
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Isthmocele
Keywords: isthmocele; cesarean section; ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- single layer: patients who underwent caesarean section with hysteroraffia performed in single layer
- double layer: patients who underwent caesarean section with double-layer hysteroraffia

SUMMARY:
The main objective of this study is to compare the frequency of isthmocele after caesarean section according to the type of hysteroraffia performed (single or double layer suture).

DETAILED DESCRIPTION:
The effects of caesarean sections on maternal health have long been known and are an issue of great interest and concern every time these epidemiological data are analysed. Among the late complications reported in the literature, several publications have analysed the correlation between the presence of abnormal uterine bleeding in the postmenstrual phase and the presence of a defect in the anterior wall of the uterine isthmus at the site of a previous caesarean section scar. Although this clinical picture, termed isthmocele, has been known for some time, its aetiopathogenesis and implications have so far been rather underestimated. The isthmocele is a saccated diverticulum of the anterior wall of the uterus in continuity with the uterine cavity, which forms at the level of the isthmus, at the site of a previous hysterectomy by caesarean section. This wall defect can lead to symptoms such as menorrhagia, abnormal uterine bleeding, pelvic pain and dysmenorrhoea. pelvic pain and dysmenorrhoea, and can also cause 'scar pregnancy' and secondary infertility. This complication occurs in more than 50% of women who undergo a caesarean section, and this percentage increases in relation to the number of previous caesarean sections. Currently, treatment options include conservative treatment, based on combined oestrogen-progestin therapy, and surgical treatment, based on hysteroscopic, laparoscopic or transvaginal repair. The choice is made on the basis of the extent of the defect, presence of symptoms, concomitant secondary infertility and desire for offspring. Although the possibility of treating isthmocele exists, in recent years interest has shifted to the possibility of preventing the occurrence of this complication. Among the risk factors recognised to date are include uterine position in retroversion and multiple caesarean sections. However, they may also contribute. However, factors such as a low uterine incision, incomplete closure of the hysterotomy, the appearance of early uterine wall adhesions and a genetic predisposition of the patient can also contribute to the development of a isthmus. A study of the risk factors associated with the occurrence of this problem showed that the technique of suturing is the most modifiable risk factor. In this regard, some studies have suggested that a double-layer closure of the uterine breach reduces the occurrence of isthmocele and increases the residual myometrial thickness, but systematic reviews of the literature have found no difference between patients undergoing single- and double-layer hysteroraffia, while they have shown that hollow sutures may lead to a larger isthmocele and a higher risk of uterine rupture, without providing any substantial haemostatic benefit. substantial haemostatic benefits. To date, there are no guidelines identifying the optimal time to perform evaluation of the cesarean section scar and diagnose the possible presence of a isthmocele. The isthmocele presents itself sonographically as a triangular anechogenic space, at least 2 mm deep, in the context of the anterior uterine wall, at the presumed site of the caesarean section scar with the base communicating with the uterine cavity. It should not be confused with the caesarean section scar itself, which appears as a hypercogenic line at the presumed site or with similar echogenicity to the surrounding myometrium. Most authors have focused on measuring the depth of the isthmocele, the size of the residual myometrial thickness and only a few have distinguished the extent of the defect into major or minor on the basis of the percentage of myometrium involved. However, other highly relevant parameters such as defect shape, volume, location, presence of multiple anechogenic areas etc. were not taken into account. The accurate measurement and description of these lesions is becoming increasingly important, for research, for the clinical assessment of gynaecological symptoms and for the planning of possible surgical treatment. For this reason, in 2019 Jordans et al. published an expert consensus 'Delphi protocol' to describe a standardised methodology for ultrasound assessment of isthmocele in patients non-pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective or emergency/emergency caesarean section at the centres involved.

Exclusion Criteria:

* Age <18 years;
* Pregnant women at the time of ultrasound assessment;
* Refusal to perform transvaginal ultrasound;
* Type of hysterorrhaphy performed during surgery not known;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients attending the Friuli Centrale University Health Authority - Obstetrics and Gynaecology of Tolmezzo
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of isthmocele | 3-4 months post cesarean section
  The main objective of this study is to compare the frequency of isthmocele after caesarean section according to the type of hysteroraffia performed (single or double layer suture).

SECONDARY OUTCOMES:
Different features of isthmocele according to type of hysteroraffia | 3-4 months post cesarean section
  To determine whether there are differences in isthmocele volume and residual myometrial thickness between patients undergoing hysteroraffia by single or double layer.
The role of anamnestic data of patients as risk factor for isthmocele | at enrollment
  Assess the impact of anamnestic data as possible risk factors for the development of isthmocele in the population considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) - SOC Clinica Ostetrica e Ginecologica Udine, Udine, Udine, Italy